CLINICAL TRIAL: NCT03335878
Title: Early Predictors of Brain Health and Development in Youth With T1DM
Brief Title: Brain Health and Development With T1DM
Acronym: NewT
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201601135
Record Dates: First submitted 2017-05-18; First posted 2017-11-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: T1DM; Brain Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participants will undergo a Mixed Meal Tolerance Test (MMTT) for assessment of residual β-cell function. A dose of Boost High Protein Nutritional Energy Drink (Mead-Johnson) mixed meal at 6 mL/kg (maximum dose 360 mL) will be given at 0 min. Blood samples will be obtained for measurement of plasma glucose and C-peptide at -10, 0, 15, 30, 60, 90, 120, 150, 180, 210, and 240 min. A split duplicate sample for quality control will be collected at either 0 or 240 min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes Mellitus Group: T1DM Group - 150 otherwise healthy children, ages 4-16 years old, diagnosed with T1DM within 3 months prior to their initial study visit. This is not a treatment study therefore there is no intervention in this study.
- Healthy Control Sibling Group: Sibling Control Group - 50 age and gender matched healthy siblings without a diagnosis of T1DM. This is not a treatment study therefore there is no intervention in this study.

SUMMARY:
Type 1 diabetes mellitus (T1DM) is typically diagnosed in childhood and over time can lead to complications affecting the retina, heart, kidneys, peripheral nerves, and more recently appreciated, the brain. Studies consistently find that early age of onset and, to a more variable extent, poor glycemic control over years are associated with reduced cognitive performance and altered brain structure in children with T1DM. As yet, the investigators' understanding of why early age of onset would pose more risks for the brain is limited, making interventions difficult to develop. Given that the initial clinical presentation of T1DM in children is the earliest and often the most severe glycemic state experienced over the lifetime, it is possible that age of onset and severity of initial clinical presentation interact to modify risks for brain health and development. This hypothesis has clear clinical implications and the potential to resolve conflicting literature, yet has not been explicitly tested. Thus, the goal of this study is to determine how clinical features at the time of T1DM diagnosis, such as hyperglycemia, diabetic ketoacidosis (DKA) and degree of beta cell failure, interact with age of onset to shape the development of the brain and its responses to subsequent glycemic control.

DETAILED DESCRIPTION:
NewT study staff will work with inpatient diabetes nurses and clinical diabetes educators at St. Louis Children's Hospital to identify patients that are admitted for new onset T1DM. Once the patients are clinically stable, the diabetes educator will visit the patient in the inpatient room and invite the family to participate in the study. If study participants would like to be enrolled, consent and assent will be obtained at that time. If potential participants are unsure at that time, the diabetes educator will provide the family with a blank copy of the consent form to be reviewed. Study information as well as contact information for study staff so that the family may contact the study should the family have additional questions or choose to enroll in the study. Following is a description of the testing days.

Mixed Meal Tolerance Tests (MMTTs) Once the patient has been consented to participate in the study, in the T1DM group, a Mixed-Meal Tolerance Tests (MMTT) will be administered at both study visits (3 mo & 21 mo post diagnosis). If participants are in the control group, the MMTT will only be administered at the 21 mo visit (18 months after the initial visit). For the MMTT, the T1DM group will be instructed to consume at least 150 g of carbohydrates per day for 3 days prior to the MMTT and to consume only water after midnight on the night prior to testing. If the patient is on insulin injection therapy the study nurse will ask the patient to administer the usual basal insulin dose(s) on the night before or on the morning of the study but to hold the morning dose of short- and intermediate-acting insulin. If the patient is on a continuous subcutaneous insulin pump infusions will remain on the usual basal rates for the duration of the study. For the MMTT a small needle, will be placed to collect blood samples. While there are multiple collection times, there is only one stick. The study nurse will then ask participants to drink a Boost High Protein Nutritional Energy Drink. Blood samples will then be obtained at the following time points: -10, 0, 15, 30, 60, 90, 120, 150, 180, 210, and 240 min. This amounts to approximately 4.5 tablespoons of blood. To clarify, only the T1DM group will have the MMTT at the first study visit (3 mo after T1DM dx), both the T1DM and the Control groups will have MMTT at the 21 month visit.

Cognitive Testing The cognitive testing or thinking tests, consist of memory tests, computer games and vocabulary tests. These tests will be administered by a trained staff member and will take approximately 60 minutes to complete. Some of the tests are: a Picture Vocabulary Test, a Picture Sequence Memory Test; an Inhibitory Control and Attention Test; a Dimensional Change Card Sort Test, and a List Sorting Working Memory Test.

Before and after the cognitive testing, blood glucose levels will be determined (using a finger prick) for participants in both groups. Participants with blood glucose values below 70 mg/dl or above 300 mg/dl will be treated and re-tested before testing resumes.

At some point during the study, one parent from each family will be requested to perform a brief reading test that provides an estimated intelligence quotient (IQ). This test takes approximately 10 minutes.

Interviews Study staff will obtain the parent/guardian's permission to access the patient's medical records in order to obtain information related to the patient's HbA1c, DKA admissions and severe hypoglycemic episodes from clinic or hospital visits. In addition, study staff will interview the proxy regarding these experiences to get additional detail that may not be captured in the records.

Questionnaires

The proxy will be asked to fill out a study questionnaire either prior to the study visit via an on-line survey or in person at the study visit. The questionnaire consists of information related to:

* For parents:

  * demographics, education and occupation,
  * behavior checklists as it pertains to the participant as well as
  * questionnaires asking about the participants' every day activity related to memory and daily functioning.
* For participants:

  * self-report behavioral information as well as
  * questionnaires asking about every day activity related to the participants' memory and daily functioning.

If at any time study participants are uncomfortable completing the questionnaire, are free to skip any questions that

Magnetic Resonance Imaging (MRI) Participants in both the T1DM and the Control groups will have an image of the brain at the 3 mo. and the 21 mo visits. An MRI is a non-invasive test to evaluate the anatomy of the different areas of the brain. A more detailed MRI than the MRI commonly used in patient care in regular hospitals is planned because we want to make specialized measurements. This test will take 45-60 minutes. No use of sedation or IV (through the vein) contrast is planned. The scan involves asking the patient to lie very still on a small table for 45-60 minutes. After the participant is comfortable on the table it will then slowly move the participant into the scanner. If the participant would like, a movie will be available to watch while in the scanner except for a short period of time when the participant will be asked to stare at a crosshair on the screen.

ELIGIBILITY:
T1DM Group

Inclusion Criteria:

* Otherwise healthy children with T1DM
* Between the ages of 4 to 16 years old
* Must be able to lie still in the MRI for 60 minutes

Exclusion Criteria:

* Mental retardation
* Enrollment in special education classes or receiving special services
* Major psychiatric (e.g. depression, autism) or neurological illnesses (e.g. head injury with loss of consciousness)
* Currently taking medications with known central nervous system effects (including those for ADHD)
* Physical limitations that would interfere with testing
* Contraindications for MRI scans
* Females who are pregnant and/or lactating will be excluded
* Chronic diseases in addition to T1DM other than well-controlled asthma, celiac disease or Hashimoto's thyroiditis as determined by their clinical endocrinologist and/or nurse

Sibling Control Group

Inclusion Criteria:

* Healthy sibling of a T1DM participant
* Matched with a T1DM participant for age and gender
* Between the ages of 4 to16 years old
* Must be able to lie still in the MRI for 60 minutes

Exclusion Criteria

* Mental retardation
* Enrollment in special education classes or receiving special services
* Major psychiatric (e.g. depression, autism) or neurological illnesses (e.g. head injury with loss of consciousness)
* Currently taking medications with known central nervous system effects (including those for ADHD)
* Physical limitations that would interfere with testing
* Contraindications for MRI scans
* Females who are pregnant and/or lactating will be excluded
* Chronic diseases other than well-controlled asthma, celiac disease or Hashimoto's thyroiditis as determined by their clinical endocrinologist and/or nurse.

The Parent population will consist of one biological parent for each minor participant. The proxy participant will complete two neuropsychological tests as well as answer questionnaires about the minor study participant. The parent population has no age limitations but must be a biological parent to the minor study participant. The testing takes approximately 20 minutes thus the parent population will not be paid for their participation.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: There are three study groups in this study.
  1. T1DM Group (n=150) Children between the ages of 4-16 yrs old who have been diagnosed with Type 1 Diabetes Mellitus (T1DM) in the past three months.
  2. Sibling Control Group (n=50) Children between the ages of 4-16 yrs old who are siblings of children with T1DM and who have NOT been diagnosed with T1DM themselves.
  3. Proxies (n=200) a parent or guardian of participants in one or both groups. The number of proxies in the study could exceed the number of minor participants because not all sibling controls have to be a sibling of a T1DM participant in the study. They may have a sibling with T1DM who doesn't meet the criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Scaled score on Verbal IQ tests at 18 months | 18 months
  The investigators hypothesize that age of onset and severity of presentation will interact to explain neuroimaging and cognitive outcomes at 3 months post-diagnosis. Specifically, the study investigators predict that patients with earlier age of onset and greater severity of clinical presentation (presence of DKA, greater HbA1c values at diagnosis) will have lower performance and more atypical brain structure and functional connectivity compared to older patients with less severe presentation and to age-matched controls, after controlling for gender, parental socioeconomic status (SES), parental IQ and intervening glycemic control. Primary neuroimaging outcomes are hippocampal volume and regional gray matter volume, microstructural white matter parameters and functional connectivity of the default mode network. Primary cognitive outcomes are memory and verbal intelligence.

SECONDARY OUTCOMES:
Functional Connectivity of the Default Mode Network at 18 months | 18 months
  The study investigators hypothesize that the development of the brain between 3 and 21 months post-diagnosis will be differently affected by severity of clinical presentation and glycemic control during follow-up. Specifically, the study investigators predict that greater severity of clinical presentation will convey greater vulnerability to subsequent hyperglycemia and severe hypoglycemia. For example, those individuals with a severe clinical presentation and significant hyperglycemia post-diagnosis will have worse outcomes on the cognitive and neuroimaging variables identified in Aim 1.
Hippocampal Volume at 18 months | 18 months
  Retrospective studies suggest that lower β-cell function uniquely predicts future long-term complications such as retinopathy, above and beyond the effects of glycemic control and duration of disease. Thus, β-cell function also may be a physiologic mediator of brain outcomes. However, prospective studies have not been conducted in newly diagnosed T1DM youth to establish that this pattern holds for the brain. Study investigators hypothesize that patients with lower β-cell function (assessed through a mixed meal tolerance test, MMTT) will be more likely to have brain and cognitive differences (identified in Aim 1) compared to those with higher β-cell function, after controlling for age, gender, parental SES, parental IQ and glycemic control.
White Matter Microstructure at 18 months | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After data is collected and entered into the REDCap database (which includes de-identifying any data) and the database is locked, the PI will then consider sharing the data with collaborators who are interested.